CLINICAL TRIAL: NCT04496284
Title: Embryo Transfer Outcomes After Vitrification With Slush Nitrogen Compared to Liquid Nitrogen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RMA-2020-03
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitrification via slush nitrogen (Experimental): Blastocyst stage embryos will be vitrified via slush nitrogen
  Interventions: Other: Vitrification via slush nitrogen
- Vitrification via liquid nitrogen (No Intervention): Blastocyst stage embryos will be vitrified via conventional liquid nitrogen. This is the current standard of care.

INTERVENTIONS:
Other: Vitrification via slush nitrogen — blastocyst stage embryos will be vitrified via slush nitrogen
  Arms: Vitrification via slush nitrogen

SUMMARY:
The proposed study is a single-blind randomized controlled trial which seeks to characterize implantation rates following embryo vitrification and subsequent warming with both slush nitrogen and liquid nitrogen. After warming, implantation rates and pregnancy outcomes will be assessed.

DETAILED DESCRIPTION:
The purpose of this study is to determine if slush nitrogen for embryo vitrification results in higher sustained implantation rates compared to the conventional use of liquid nitrogen. Routine ovarian stimulation, oocyte retrieval and embryology care will ensue. All blastocyst stage embryos will be randomized to either the control (liquid nitrogen) or intervention group (slush nitrogen) and vitrified after trophectoderm biopsy has been performed for PGT-A (preimplantation genetic testing for aneuploidy). A single, chromosomally normal embryo will be transferred in a subsequent frozen embryo transfer cycle per routine. Implantation rates and pregnancy outcomes will be assessed.

ELIGIBILITY:
Major Inclusion Criteria for participants:

1. Patients undergoing IVF stimulation cycle with plan for subsequent frozen embryo transfer (FET)
2. Patients electing preimplantation genetic testing for aneuploidy (PGT-A)
3. Couples electing single embryo transfer (SET)

Major Exclusion Criteria for participants:

1. All patients who do not voluntarily give their written consent for participation
2. Under 18 years old, above 42 years old
3. BMI > 35
4. Maximum day 3 Follicle stimulating hormone (FSH) level of 12 or higher
5. Anti-mullerian hormone (AMH) level less than 1.0 g/mL, tested within previous year
6. Total basal antral follicle count less than 6 follicles
7. Failed more than one previous FET cycle
8. Use of oocyte donation
9. Use of gestational carrier
10. Presence of hydrosalpinges that communicate with endometrial cavity
11. Diagnosis of endometrial insufficiency: prior cycle with maximal endometrial thickness ≤ 6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), persistent endometrial fluid
12. Uncorrected uterine factor infertility (uterine anomaly, submucosal myomas, uterine septum)
13. Single gene disorder chromosomal rearrangement requiring a more detailed embryonic genetic analysis
14. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
15. Use of surgical procedures to obtain sperm
16. Couples undergoing IVF for fertility preservation with no immediate plan for subsequent FET (embryo banking)
17. Sex selection
18. Personal history of repeated pregnancy loss (two or more unexplained clinical losses defined by presence of fetal heartbeat)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
sustained implantation rate | approximately 8 weeks gestation age
  fetal heart beat present upon discharge at 8 weeks

SECONDARY OUTCOMES:
clinical pregnancy rate | usually by 5 weeks gestational age
  presence of gestational sac in uterus
miscarriage rate | 1-8 months dependent on gestational age of loss
  pregnancy loss
live birth rate | 9 months
  delivery of live infant

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klimczak AM, Osman E, Esbert M, Yildirim RM, Whitehead C, Herlihy NS, Hanson BM, Roberts LM, Seli E, Scott RT Jr. A randomized controlled trial comparing embryo vitrification with slush nitrogen to liquid nitrogen in women undergoing frozen embryo transfer: embryology and clinical outcomes. Hum Reprod. 2025 Mar 1;40(3):426-433. doi: 10.1093/humrep/deaf003. PMID 39836897